CLINICAL TRIAL: NCT06598670
Title: Effects of Transcranial Direct Current Stimulation on Post Stroke Depression
Brief Title: Transcranial Direct Current Stimulation on Post Stroke Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC02030 Jaweria Zaib Abbasi
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Post-stroke Depression
Keywords: Stroke; depression; transcranial direct current stimulation
MeSH Terms: conditions — Stroke; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS Group (Experimental): Active tDCS will be applied to the M1 area of the brain with the conventional therapy
  Interventions: Other: tDCS; Other: Conventional treatment
- Sham tDCS Group (Active Comparator): Sham tDCS will be applied to the M1 area of the brain with the conventional therapy
  Interventions: Other: tDCS; Other: Conventional treatment

INTERVENTIONS:
Other: tDCS — tDCS will be applied to the M1 area for 20 minutes with 5x7 cm electrodes. The intervention will be applied for eight weeks on alternate days
Other: Conventional treatment — Breathing exercises will be performed

SUMMARY:
The aim of the research is to address the critical gap that limited number of RCTs are conducted on this topic. To further explore the efficacy of tDCs, large sample sizes, large follow up period and rigorously controlled randomized clinical trials are necessary. An optimum stimulation protocol is also needed on this study. Previous studies lack information regarding effects of this stimulation on depression, cognition, quality of life in relation to different severity levels of stroke.

DETAILED DESCRIPTION:
Research studies revealed that PSD causes both cognitive and physical impairments to lower motivation, which hinders rehabilitation program participation and slows down executive functions. Due to depression, cognitive dysfunctions difficulty in executive, working memory and emotional deficits which declines quality of life (QoL). Thus, the combined effects of cognitive decline and PSD considerably more worsen stroke survivors' QoL with regard to psychological, environmental and physical well-being Evidence supports various techniques for minimizing PSD, restoring cognitive function, and enhancing QoL including mindfulness-based therapies, exercise therapy (aerobic and resistance trainings), progressive muscle relaxation exercises, cognitive behavioral therapy (CBT). Non-invasive brain stimulation (NIBS) include transcranial direct current stimulations (tDCS) demonstrated significant therapeutic outcomes in the PSD rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Stroke for more than 6 months Both gender with equal ratio on stroke severity basis Depression diagnosed by Psychiatrist Mild and moderate Depression at PHQ-9 National Institutes of Health Stroke Scale (NIHSS) for severity level; Mild (1-4), Moderate (5-15), Moderate to Severe (16-20), Severe (21-42)

Exclusion Criteria:

* Any medical condition like cardiac arrhythmias, uncontrolled hypertension. Individual with any pacemaker and metal implant in body. Patient with any other neurological and psychiatric condition.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) for depression | 8 weeks
  Patient Health Questionnaire (PHQ-9) is a self-administered and widely used tool for screening, diagnosing, monitoring, and measuring post stroke depression .It consists of 9 items, scored from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. The PHQ-9 interpreted as 0-4=No depression, 5-9=mild depression, 10-14=Moderate depression, 15- 19=Moderately severe, 20-27=severe depression.
MoCA | 8 weeks
  Montreal Cognitive Assessment (MoCA) plays a significant role in the prediction of Cognitive Impairment after stroke. MoCA is scored out of 30 points. Interpreted as 26-30=Normal Cognitive impairment 18-25 = mild cognitive impairment, 10-17= moderate cognitive impairment and less than 10= severe cognitive impairment.

SECONDARY OUTCOMES:
SS-QoL | 8 weeks
  SS-QOL is a tool designed for self-assessment of stroke survivors. It might be completed by the patient or its caregiver, as the time required to complete is 10-15 minutes. The questionnaire consists of 49 items divided in 12 domains; energy, family role, language, mobility, mood, personality, self-care, social role, thinking, upper extremity function, vision and work. Five-point Likert scale. The results are later rescaled to fit the 0 to100 scale where 100 is being the best health state.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chohan SA, Venkatesh PK, How CH. Long-term complications of stroke and secondary prevention: an overview for primary care physicians. Singapore Med J. 2019 Dec;60(12):616-620. doi: 10.11622/smedj.2019158. PMID 31889205
- [Background] Sarkar A, Sarmah D, Datta A, Kaur H, Jagtap P, Raut S, Shah B, Singh U, Baidya F, Bohra M, Kalia K, Borah A, Wang X, Dave KR, Yavagal DR, Bhattacharya P. Post-stroke depression: Chaos to exposition. Brain Res Bull. 2021 Mar;168:74-88. doi: 10.1016/j.brainresbull.2020.12.012. Epub 2020 Dec 31. PMID 33359639
- [Background] Zhou L, Wang L, Liu G, Cai E. Prognosis prediction models for post-stroke depression: a protocol for systematic review, meta-analysis, and critical appraisal. Syst Rev. 2024 May 22;13(1):138. doi: 10.1186/s13643-024-02544-x. PMID 38778417
- [Background] Hao W, Liu Y, Gao Y, Gong X, Ning Y. Transcranial direct current stimulation for the treatment of post-stroke depression: A systematic review. Front Neurol. 2023 Jan 18;13:955209. doi: 10.3389/fneur.2022.955209. eCollection 2022. PMID 36742053
- [Background] Herrera-Melendez AL, Bajbouj M, Aust S. Application of Transcranial Direct Current Stimulation in Psychiatry. Neuropsychobiology. 2020;79(6):372-383. doi: 10.1159/000501227. Epub 2019 Jul 24. PMID 31340213